CLINICAL TRIAL: NCT01182012
Title: Reduction of Cardiovascular Risk in Severe Mental Illness Prescribing and Using Better and More Appropriated Drugs
Brief Title: Reduction of Cardiovascular Risk in Severe Mental Illness
Acronym: RISCA-TMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Hospitalari de Vic (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Quintí Foguet-Boreu, MD & PhD, Vic Hospital Consortium - Consorci Hospitalari de Vic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CVD-SMI-2009-03
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Severe Mental Illness; Schizophrenia; Bipolar Disorder; Affective Disorders; Schizoaffective Disorder; Personality Disorder
Keywords: Cardiovascular risk factor; Severe mental illness; Drug appropriateness; Drug compliance; Lifestyle counseling
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Mood Disorders; Psychotic Disorders; Personality Disorders; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): Adjust drug treatment to control cardiovascular factor risks. A nurse will implement a lifestyle counseling in order to improve compliance of treatment and a healthy lifestyle.
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — Depending on the results of cardiovascular risk factor indexes, the treatment (including drugs, if needed) may be modified or adjusted. A nurse visit will be programmed to explain the lifestyle behaviour the patient should have.

SUMMARY:
Background:

Patients with severe mental illness (SMI) have a higher prevalence of cardiovascular risk factors (CVRF) than the general population and a control of these risk factors poorer. Serious mental illness often causes health teams to focus interventions in mental illness and put aside the CVRF.

Objectives:

This project aims to assess the CVRF, stratify the cardiovascular risk, adequate drug treatment to reduce this risk and evaluate the effectiveness of an intervention by professional community nurses in patients with SMI.

Materials and Methods:

Prospective study of a cohort of patients over 18 years with a diagnosis of SMI with two cross sections to evaluate the cardiovascular risk and adequacy of drug treatment. The investigators calculate the risk to the cardiovascular risk tables with the SCORE (Systematic Coronary Risk Evaluation) for countries of low cardiovascular risk and the of Framingham REGICOR (Heart registry of Girona, Spain). The adequacy of pharmacotherapy will be assessed contrasting it with the recommendations of the Program of Preventive Activities and Health Promotion of Family medical association. The intervention will be conducted by professional nurses and consist of an initial psycho-educational intervention, and two more reinforcement throughout twelve months, of duration less than 30 minutes that will be addressed in an integrated manner the clinical situation with regard to cardiovascular risk. If necessary, pharmacological treatment will be prescribed. Twelve months after the first intervention, a second evaluation on cardiovascular risk and the effectiveness of the intervention will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a severe mental illness as schizophrenia, bipolar disorder, affective disorder, schizoaffective disorder or personality disorder and others who receive clinical follow-up in Osona (a county) mental health center.
* Inclusion will be delayed in patients with acute psychiatric symptoms.

Exclusion Criteria:

* Renal or hepatic failure, metabolic or endocrine disorder
* Patients who do not accept to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of cardiovascular risk | After one year of inclusion
  To collect the Systematic coronary risk evaluation (SCORE) index adapted for low-risk countries and the REGICOR index (an adaptation on the Framingham cardiovascular risk function) for each patient twice at inclusion and after one year of follow-up. To calculate and to analyse the changes between the two moments.

SECONDARY OUTCOMES:
Normalization of blood pressure | After one year of inclusion
  An analysis will be made to see if initial abnormal blood pressure levels have been normalized at the end of study.
Normalization of cholesterolemia | After one year of inclusion
  An analysis will be made to see if initial abnormal cholesterolemia blood levels have been normalized at the end of study.
Control of hiperglycaemia | After one year of inclusion
  An analysis will be made to see if initial abnormal glycose blood levels (and if diabetes was diagnosticated) have been normalized at the end of study.
Smoking cessation | After one year of inclusion
  At the end of follow-up an study about smoking cessation will be made.
Euro-Qol index | After one year of inclusion
  To compare Euro-Qol index quality of life questionnaire obtained twice, at inclusion and after one year of follow-up.
Seville quality of life questionnaire (SQLQ) | After one year of inclusion
  Seville quality of life questionnaire has proven to be a valid sensitive instrument to measure quality of life in schizophrenic patients. It focuses on aspects that are relevant for patients that were frequently overlooked by treating physicians. To compare SQLQ index obtained twice, at inclusion and after one year of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Quintí Foguet-Boreu, MD, PhD, Principal Investigator — Vic Hospital Consortium - Consorci Hospitalari de Vic
Locations (1):
- Vic Hospital Consortium - Consorci Hospitalari de Vic, Vic, Catalonia, Spain

REFERENCES:
- [Background] Hayward C. Psychiatric illness and cardiovascular disease risk. Epidemiol Rev. 1995;17(1):129-38. doi: 10.1093/oxfordjournals.epirev.a036169. PMID 8521931
- [Background] Gold KJ, Kilbourne AM, Valenstein M. Primary care of patients with serious mental illness: your chance to make a difference. J Fam Pract. 2008 Aug;57(8):515-25. No abstract available. PMID 18687227
- [Background] Maj M. Physical health care in persons with severe mental illness: a public health and ethical priority. World Psychiatry. 2009 Feb;8(1):1-2. doi: 10.1002/j.2051-5545.2009.tb00196.x. No abstract available. PMID 19293947
- [Background] Heald A, Montejo AL, Millar H, De Hert M, McCrae J, Correll CU. Management of physical health in patients with schizophrenia: practical recommendations. Eur Psychiatry. 2010 Jun;25 Suppl 2:S41-5. doi: 10.1016/S0924-9338(10)71706-5. PMID 20620887
- [Background] Marrugat J, Solanas P, D'Agostino R, Sullivan L, Ordovas J, Cordon F, Ramos R, Sala J, Masia R, Rohlfs I, Elosua R, Kannel WB. [Coronary risk estimation in Spain using a calibrated Framingham function]. Rev Esp Cardiol. 2003 Mar;56(3):253-61. doi: 10.1016/s0300-8932(03)76861-4. Spanish. PMID 12622955
- See also: Cardiovascular risk in severe mental illness — http://www.chv.cat